CLINICAL TRIAL: NCT05499728
Title: Physical Therapy Following Shoulder Arthroplasty: An Assessment of Telerehabilitation vs. In-Person Physical Therapy
Brief Title: Telerehabilitation After Shoulder Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brendan M. Patterson, Physician, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202104097
Record Dates: First submitted 2022-07-15; First posted 2022-08-12 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Arthritis Shoulder Glenohumoral Joint; Rotator Cuff Tear Arthropathy; Arthropathy Shoulder
Keywords: Shoulder arthroplasty; Physical therapy; Telerehabilitation
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Subjects who are randomized to telerehabilitation will be provided access to telemedicine visits with a physical therapist. Patients will have one in-person physical therapy visit before starting telerehabilitation, and another in-person visit at 3 months to assess progress. Telerehabilitation visits will be performed via secure usage of the electronic medical record (EMR). To ensure uniformity, and to allow for appropriate access to telehealth services, all telehealth visits will be carried out through the study institution's Department of Physical Therapy. It is expected most patients will complete formal physical therapy by 6 months postoperative measured by the time at which patient's regain functional range of motion or patients are satisfied with their results. Shoulder range of motion will be measured with a goniometer preoperatively, as well as 3,6, 12, and 24 months postoperatively at their regularly scheduled clinic visit.
  Interventions: Other: Telerehabilitation; physical therapy via telecommunication device (i.e. online video conferencing)
- Traditional In-Person Physical Therapy (No Intervention): Subjects who are randomized to in-person therapy will present to a physical therapist of their choice with a established written protocol. The therapy protocol is developed in conjunction with the Department of Orthopaedic Surgery and the Department of Physical Therapy. Subjects are recommended to attend in-person appointments at least once a week as well as perform home exercises. Progress with therapy will be collected with weekly phone calls from the research team. It is expected most subjects will complete formal physical therapy by 6 months postoperative attending on average 5-6 visits, measured by the time at which patient's regain functional range of motion or are instructed by their therapist to discontinue. Shoulder range of motion will be measured with a goniometer preoperatively, as well as 3,6, 12, and 24 months postoperatively at their regularly scheduled clinic visit.

INTERVENTIONS:
Other: Telerehabilitation; physical therapy via telecommunication device (i.e. online video conferencing) — Postoperative physical therapy performed through online video conferencing with a licensed physical therapist while the patient remains remote/at home rather than in person
  Arms: Telerehabilitation

SUMMARY:
The use of reverse total shoulder arthroplasty (RSA) has increased dramatically in the United States in recent years. The importance of postoperative physical therapy in the setting of anatomic total shoulder is well understood and explored in the literature. The literature describing postoperative physical therapy for RSA, however, is scarce and somewhat limited to the field of physiatry in the form of clinical commentary on rehabilitation programs.In addition, the use of formal in-person therapy versus physician-guided home therapy has been explored in total shoulder arthroplasty, demonstrating similar post-operative range of motion and patient-reported outcome (PROs) between groups. Furthermore, previous research into "telerehabilitation" or remote physical therapy through a video-based platform has demonstrated noninferiority in outcomes in multiple orthopedic procedures, including hip and knee arthroplasty and reverse shoulder arthroplasty. Telehealth therapy has not yet been formally evaluated in a randomized approach for reverse or anatomic total shoulder arthroplasty. Given the ongoing COVID-19 pandemic, emphasis on social distancing, and multiple states having issued "stay at home" orders, a study into the effectiveness of telerehabilitation on current postoperative outcomes in shoulder arthroplasty may influence postoperative management and allow patients an alternative route for rehabilitation that allows more flexibility in completing, as well as limits potentially extraneous travel and exposure. The project will be a randomized control trial evaluating formal in-person physical therapy versus telerehabilitation after shoulder arthroplasty. Patients who undergo shoulder arthroplasty will complete either formal physical therapy or telerehabilitation postoperatively. The aim will be to identify any differences in shoulder range of motion, pain, or patient-reported outcome measures (PROs) between those who complete in-person physical therapy versus telerehabilitation therapy.

DETAILED DESCRIPTION:
After agreeing to participate and signing the informed consent, subjects will be randomized into in person physical therapy group or telerehabilitation group. At the 2-week postoperative visit, the subject will receive a sealed envelope which will contain the information about the group they have randomly been assigned to. Both groups (in person therapy and telerehabilitation) are expected to start physical therapy at 6-week after surgery, this means that all subjects will have 4 weeks after being assigned to program and organize for physical therapy.

Subjects who are randomized to in-person therapy will present to a physical therapist of their choice with a established written protocol. The therapy protocol is developed in conjunction with the Department of Orthopaedic Surgery and the Department of Physical Therapy. Subjects are recommended to attend in-person appointments at least once a week as well as perform home exercises. Progress with therapy will be collected with weekly phone calls from the research team. It is expected most subjects will complete formal physical therapy by 6 months postoperative attending on average 5-6 visits, measured by the time at which patient's regain functional range of motion or are instructed by their therapist to discontinue. Shoulder range of motion will be measured with a goniometer preoperatively, as well as 3,6, 12, and 24 months postoperatively at their regularly scheduled clinic visit. (Shoulder arthroplasty patients regularly return to clinic at these intervals and would not be required to present to clinic in addition to these time points. Patients also regularly return to clinic at 2 weeks and 6 weeks postoperatively as a part of their normal clinical follow up for wound check and general assessment.) Subjects who are randomized to telerehabilitation will be provided access to telemedicine visits with a physical therapist. These patients will have one first in-person physical therapy visit before starting telerehabilitation, and another in-person physical therapy visit at 3 months to assess progress. Telerehabilitation visits will be performed via secure usage of the electronic medical record (EMR). Progress with telerehabilitation will be collected with weekly phone calls from the research team. To ensure uniformity, and to allow for appropriate access to telehealth services, all telehealth visits will be carried out through the study institution's Department of Physical Therapy. It is expected most patients will complete formal physical therapy by 6 months postoperative measured by the time at which patient's regain functional range of motion or patients are satisfied with their results. Shoulder range of motion will be measured with a goniometer preoperatively, as well as 3,6, 12, and 24 months postoperatively at their regularly scheduled clinic visit. (Shoulder arthroplasty patients regularly return to clinic at these intervals and would not be required to present to clinic in addition to these time points. Patients also regularly return to clinic at 2 weeks and 6 weeks postoperatively as a part of their normal clinical follow up for wound check and general assessment.)

Review of the medical record will collect the following demographic information: medical record number, surgical date, age, BMI, smoking status, rheumatoid arthritis diagnosis, rotator cuff arthropathy diagnosis, subscapularis repair description, intraoperative integrity of the rotator cuff, physical therapy modality (in-person vs. telerehabilitation), physical therapy progress notes, and therapy compliance. Outcome measures will include shoulder range of motion including forward flexion, internal and external rotation, and all patient-reported outcome measures (PROs) assigned to shoulder arthroplasty patients already available for collection in Epic.

ELIGIBILITY:
Inclusion Criteria:

* All patients being indicated for primary shoulder arthroplasty, both anatomic and reverse shoulder arthroplasty, by one of two orthopedic shoulder surgeons.

Exclusion Criteria:

* Patients undergoing revision procedures, concomitant procedures (for example, tendon transfer), arthroplasty for fracture, and those who do not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder range of motion | 2 years
  Patient's ability to actively and passively move the shoulder in multiple planes of motion
American Shoulder and Elbow Surgeons score | 2 years
  A patient reported outcome measure utilizing a 100-point scale that assesses pain (50 points) and activities of daily living (50 points). A higher score (100) indicates a better shoulder condition.
PROMIS Pain Interference | 2 years
  A patient reported outcome measure detailing self-reported consequences of pain and the extent to which, over a immediate 7-day recall period, pain influences patient well-being and activity. A higher score indicates a higher degree of pain interference.
PROMIS Global Health score | 2 years
  A patient reported outcome measure detailing self-reported markers of overall patient health. A higher score represents a healthier patient in that specific domain.
Visual Analog Scale for Pain | 2 years
  A patient reported outcome measure detailing pain intensity using a numerical value from 1-10. A higher score indicates worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia O'Reilly, MD, Principal Investigator — University of Iowa; Brendan M Patterson, MD, MPH, Principal Investigator — University of Iowa
Locations (1):
- Brendan Patterson, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palsis JA, Simpson KN, Matthews JH, Traven S, Eichinger JK, Friedman RJ. Current Trends in the Use of Shoulder Arthroplasty in the United States. Orthopedics. 2018 May 1;41(3):e416-e423. doi: 10.3928/01477447-20180409-05. Epub 2018 Apr 16. PMID 29658976
- [Background] Chalmers PN, Salazar DH, Romeo AA, Keener JD, Yamaguchi K, Chamberlain AM. Comparative Utilization of Reverse and Anatomic Total Shoulder Arthroplasty: A Comprehensive Analysis of a High-volume Center. J Am Acad Orthop Surg. 2018 Dec 15;26(24):e504-e510. doi: 10.5435/JAAOS-D-17-00075. PMID 30161057
- [Background] Wright MA, Keener JD, Chamberlain AM. Comparison of Clinical Outcomes After Anatomic Total Shoulder Arthroplasty and Reverse Shoulder Arthroplasty in Patients 70 Years and Older With Glenohumeral Osteoarthritis and an Intact Rotator Cuff. J Am Acad Orthop Surg. 2020 Mar 1;28(5):e222-e229. doi: 10.5435/JAAOS-D-19-00166. PMID 31356423
- [Background] Bullock GS, Garrigues GE, Ledbetter L, Kennedy J. A Systematic Review of Proposed Rehabilitation Guidelines Following Anatomic and Reverse Shoulder Arthroplasty. J Orthop Sports Phys Ther. 2019 May;49(5):337-346. doi: 10.2519/jospt.2019.8616. Epub 2019 Apr 25. PMID 31021690
- [Background] Mulieri PJ, Holcomb JO, Dunning P, Pliner M, Bogle RK, Pupello D, Frankle MA. Is a formal physical therapy program necessary after total shoulder arthroplasty for osteoarthritis? J Shoulder Elbow Surg. 2010 Jun;19(4):570-9. doi: 10.1016/j.jse.2009.07.012. Epub 2009 Oct 2. PMID 19800258
- [Background] Keener JD, Galatz LM, Stobbs-Cucchi G, Patton R, Yamaguchi K. Rehabilitation following arthroscopic rotator cuff repair: a prospective randomized trial of immobilization compared with early motion. J Bone Joint Surg Am. 2014 Jan 1;96(1):11-9. doi: 10.2106/JBJS.M.00034. PMID 24382719
- [Background] Boudreau S, Boudreau ED, Higgins LD, Wilcox RB 3rd. Rehabilitation following reverse total shoulder arthroplasty. J Orthop Sports Phys Ther. 2007 Dec;37(12):734-43. doi: 10.2519/jospt.2007.2562. Epub 2007 Aug 28. PMID 18560182
- [Background] Uschok S, Herrmann S, Pauly S, Perka C, Greiner S. Reverse shoulder arthroplasty: the role of physical therapy on the clinical outcome in the mid-term to long-term follow-up. Arch Orthop Trauma Surg. 2018 Dec;138(12):1647-1652. doi: 10.1007/s00402-018-3015-9. Epub 2018 Jul 30. PMID 30062455
- [Background] Romano AM, Oliva F, Nastrucci G, Casillo P, Di Giunta A, Susanna M, Ascione F. Reverse shoulder arthroplasty patient personalized rehabilitation protocol. Preliminary results according to prognostic groups. Muscles Ligaments Tendons J. 2017 Sep 18;7(2):263-270. doi: 10.11138/mltj/2017.7.2.263. eCollection 2017 Apr-Jun. PMID 29264337
- [Background] Wolff AL, Rosenzweig L. Anatomical and biomechanical framework for shoulder arthroplasty rehabilitation. J Hand Ther. 2017 Apr-Jun;30(2):167-174. doi: 10.1016/j.jht.2017.05.009. PMID 28641735
- [Background] Simovitch R, Flurin PH, Wright T, Zuckerman JD, Roche CP. Quantifying success after total shoulder arthroplasty: the minimal clinically important difference. J Shoulder Elbow Surg. 2018 Feb;27(2):298-305. doi: 10.1016/j.jse.2017.09.013. Epub 2017 Nov 20. PMID 29162305
- [Background] Wagner ER, Solberg MJ, Higgins LD. The Utilization of Formal Physical Therapy After Shoulder Arthroplasty. J Orthop Sports Phys Ther. 2018 Nov;48(11):856-863. doi: 10.2519/jospt.2018.8176. Epub 2018 May 8. PMID 29739303
- [Background] Palm KB, Blazar PE, Manna JC, Serig AS, Phillips EA, Bay CP, Casey EJ, Earp BE. Feasibility, effectiveness and patient satisfaction of telerehabilitation after thumb carpometacarpal arthroplasty and reverse total shoulder arthroplasty: A pilot study. J Telemed Telecare. 2023 Aug;29(7):521-529. doi: 10.1177/1357633X21999578. Epub 2021 Mar 5. PMID 33673751
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Estebanez-Perez MJ. Evidence of Benefit of Telerehabitation After Orthopedic Surgery: A Systematic Review. J Med Internet Res. 2017 Apr 28;19(4):e142. doi: 10.2196/jmir.6836. PMID 28455277